CLINICAL TRIAL: NCT02990754
Title: Fearless Physical Activity: Getting and Keeping Ontarians With Congenital Heart Disease Active in Community Sport, Recreation and Physical Activity
Brief Title: Fearless Physical Activity: Getting and Keeping Ontarians With Congenital Heart Disease Active
Acronym: Fearless
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Congenital Heart Alliance (Other)
Responsible Party: Principal Investigator, Dr. Pat Longmuir, Scientist, Children's Hospital of Eastern Ontario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16/106X
Record Dates: First submitted 2016-12-06; First posted 2016-12-13 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Group (Experimental): Individuals attending one or more fearless physical activity events
  Interventions: Behavioral: Physical activity education

INTERVENTIONS:
Behavioral: Physical activity education — Instruction in suitable physical activity options and education about physical activity with CHD.

SUMMARY:
"Fearless Physical Activity" are fun, physical literacy events where people with congenital heart disease (CHD) and sport/recreation leaders can do community-based sport/recreation opportunities "without fear" (i.e., appropriate for their health). Ontarians with CHD are a large and rapidly growing population;1% of children are born with CHD, adding 1,440 new children/year to the 113,900 Ontarians of all ages who are living with CHD. 'Fearless' will target CHD children, youth or adults, while encouraging family-based participation. During each season, the investigators will offer a one-day event for each age group (children, youth, adults) in each region of Ontario (4 seasons x 3 age groups x 4 regions = 48 events). Event activities will be hosted by community partners, such as the MLSE Launch Pad (Toronto) or the YMCA/YWCA of the National Capital Region (Ottawa), so that they are sustainable beyond this project. Activities will be chosen based on opportunities available in local communities at little to no cost (e.g., use of local trails and parks). Event leaders and participants will be educated about physical literacy and screening tasks will be used to identify those needing significant or specialized physical literacy support. People with CHD lead mostly sedentary lives. They are much less active than their friends and colleagues, even when their heart disease is mild, and inactivity can contribute to a higher risk for heart attacks, stroke, obesity, and depression. Uncertainty about physical activity, even though it is recommended (American Heart Association, May 2014), is an important barrier to the physical and mental health benefits of physical activity. "How much is too much?" and "Will it be too much for my heart?" are top-of-mind. "Fearless Physical Activity" will provide children, youth and adults living with CHD with new physical activity experiences and opportunities to enhance their physical literacy so they are better able to be "active for life".

DETAILED DESCRIPTION:
"Fearless Physical Activity" will deliver high-quality, meaningful physical literacy-enhancing experiences to children, youth and adults with congenital heart disease (CHD). People with CHD have historically been much less active than other Ontarians, regardless of heart disease severity. 'Fearless' will increase opportunities for sport/recreation participation by directly providing 48 days of fun, physical activity specifically designed for children, youth and adults with CHD and their families. Each event day, physical literacy screening tasks will identify those with CHD who are likely to require very significant support to be "active for life". 'Fearless' participants and leaders will learn about physical literacy, and it's fundamental role as the foundation of a healthy active lifestyle. A physical literacy workshop will educate leaders within the Canadian Congenital Heart Alliance (CCHA) about the importance of physical literacy for people with CHD and the role that CCHA can play in supporting active lifestyles. Joint organization of 'Fearless' events will develop new partnerships between the CCHA and the community sport and recreation sector. These partnerships will enhance sport and recreation sector capacity to understand, and better support, the physical literacy needs of people with CHD. The project outcomes will be increased physical literacy among children, youth and adults with CHD, more physically active people with CHD and enhanced sport and recreation sector capacity to provide opportunities that are accessible to Ontarians with CHD.

The planning and partnership phase of 'Fearless' (April to December 2016) will lay the groundwork for the delivery of the "Fearless Physical Activity" events. The Project Coordinator will work collaboratively with the leadership of the Canadian Congenital Heart Alliance (CCHA) and existing CCHA chapters in London and Eastern Ontario to develop the educational content and desired physical activity opportunities that will be delivered through the 'Fearless' events. A previous one-day 'Fearless' event evaluated the feasibility of our concept and the interest among families of those with CHD. The previous one-day event combined education sessions about physical activity goal setting, identifying personal activity interests, and finding community physical activity opportunities with opportunities to participate in a wide variety of physical activities (e.g., geocaching, Frisbee golf, croquet, beachball volleyball). Feedback from participating families rated all aspects of the 'Fearless' event as excellent or outstanding. However, this one event was held for children with CHD and their families during the summer, therefore the project coordinator and project partners will need to develop additional content and activity plans to ensure that we can provide events for three age groups (children, youth, adults) and in all four seasons of the year. Providing events in all four seasons is important because people with CHD are highly susceptible to temperature extremes (cold, hot) and humidity; leading many people with CHD to believe that physical activity is not a feasible option at many times of the year. During the planning phase, the project coordinator will strengthen existing partnerships and networks within the CCHA and the sport and recreation sector, as well as develop the new partnerships (recreation/sport partners in western and northern Ontario) and expanded networks (northern Ontario) needed to ensure that people with CHD know about the Fearless events, which will be offered in all regions of Ontario.

The 'Fearless' events will be held during 2017 (winter, spring, summer, fall) in each region of Ontario. Each one-day event will be held on a weekend, to facilitate the participation of people with CHD and their families. Having a series of education and activity sessions on one day, rather than shorter sessions held more frequently, will better enable people with CHD to attend from across the wide geographic areas served by each CCHA chapter / CHD clinic. Each 'Fearless' event will include education sessions, participatory physical activity opportunities and the completion of physical literacy screening tasks that will identify those needing the greatest support to be active for life. The topic for one education session will be physical literacy - its importance, how it can be developed throughout life, and its relationship to physical and mental health. Each 'Fearless' event will be hosted by a community sport and recreation partner, enhancing project sustainability and sector capacity to support the physical activity of people with CHD.

ELIGIBILITY:
Inclusion Criteria:

* child, adolescent or adult diagnosed with a congenital heart defect and their family members

Exclusion Criteria:

* disabilities that prevent the individual from safely participating in group events

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Habitual Activity Estimation Scale | 1-month post intervention
  Change from baseline in self-reported physical activity participation questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Longmuir, PhD, Principal Investigator — Scientist
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No